CLINICAL TRIAL: NCT06368778
Title: The Impact of Real-Time Biofeedback on Partial Weightbearing Training: A Comparative Study
Brief Title: Real-Time Biofeedback on Partial Weightbearing Training
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Justin Haller, Principle Investigator, University of Utah
Other Study IDs: 166591
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Physical Therapy
Keywords: Biofeedback; Loadsol device; Partial weightbearing training; Standard of care training; Healthy subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1 "Verbal Advice": The participant will receive verbal instructions following the standard of care physical therapy. A member of the study team will observe and provide comments on the participant's exercises.
  Interventions: Other: Verbal Advice
- Group 2 "Bathroom Scale": In this group, the participant is given a sense of what a 20 kg load feels like using a scale. Subsequently, the same exercises as in Group 1 will be conducted.
  Interventions: Other: Bathroom Scale
- Group 3 "Biofeedback": In this group, the biofeedback function of the sensor insoles is activated. This feature provides both visual (a bar graph on the iPad) and auditory feedback (an audible signal when the load exceeds 20 kg). Through this feedback, the participant is expected to develop an understanding of partial weight-bearing.
  Interventions: Device: Loadsol Biofeedback

INTERVENTIONS:
Other: Verbal Advice — The participant will receive verbal instructions following the standard physical therapy.
  Other Names: Standard physical therapy
  Groups: Group 1 "Verbal Advice"
Other: Bathroom Scale — The participant is given a sense of what a 20 kg load feels like using a scale.
  Other Names: 20 kg load input with standard physical therapy.
  Groups: Group 2 "Bathroom Scale"
Device: Loadsol Biofeedback — Average peak force (N) with be measured during partial weightbearing physical therapy routine for 2-minutes using the Loadsol device.
  Other Names: Loadsol device
  Groups: Group 3 "Biofeedback"

SUMMARY:
The purpose of this study is to investigate the effectiveness of a biofeedback device (Loadsol) in training healthy subjects to comply with partial weightbearing, and to compare its outcomes with the standard of care training. Partial weightbearing is an essential component of rehabilitation and recovery for many orthopedic patients, yet it remains challenging for individuals to accurately gauge their weightbearing restrictions without proper guidance and feedback.

The primary objective of the study is to determine whether the use of the biofeedback device (Loadsol) can reduce the time it takes for healthy subjects to learn and comply with partial weightbearing, compared to traditional training methods. The Loadsol device provides real-time auditory feedback on the individual's weightbearing status, potentially enhancing the learning process and adherence to weightbearing restrictions.

Secondary objectives of the study include:

Assessing the compliance of subjects with weightbearing restrictions in both the biofeedback and standard of care training groups, and comparing the results to identify any significant differences in adherence to the prescribed weightbearing limitations.

Evaluating subject satisfaction with the training methods, as measured through questionnaires and the use of Patient-Reported Outcomes Measurement Information System (PROMIS) tools. This evaluation will help determine if the biofeedback device (Loadsol) leads to higher levels of satisfaction among subjects compared to the standard of care training.

By examining these objectives, this study aims to provide valuable insights into the potential benefits of using a biofeedback device in partial weightbearing training, and to establish whether its implementation can lead to improved outcomes in learning, compliance, and overall patient satisfaction.

DETAILED DESCRIPTION:
Partial weightbearing is an essential aspect of rehabilitation for many orthopedic patients, as it promotes healing and helps prevent complications after injury or surgery. Traditionally, patients receive instructions and guidance from healthcare professionals to achieve appropriate weightbearing levels. However, accurately gauging one's weightbearing status can be challenging without proper feedback.

Recent literature has investigated the use of biofeedback devices in training patients for partial weightbearing, demonstrating their potential in improving compliance and learning. However, to date, no studies have directly compared the effectiveness of biofeedback devices, such as Loadsol, with the standard of care (SOC) in terms of the time required for patients to learn and comply with partial weightbearing restrictions.

Furthermore, existing research has focused on orthopedic patients, who may be subject to various confounding factors such as pain, different fracture patterns, and surgical interventions. No studies have yet explored the use of biofeedback devices in training healthy subjects for partial weightbearing, which could provide valuable insights without the influence of these confounders.

In addition, the Loadsol device has been compared to other devices, such as treadmills and force plates, in terms of measurement quality. Studies have suggested that the Loadsol device provides comparable results, supporting its reliability and potential effectiveness in partial weightbearing training.

This study aims to fill the gap in the literature by comparing the Loadsol biofeedback device with the standard of care in training healthy subjects for partial weightbearing. By evaluating the time taken to learn and comply with weightbearing restrictions, compliance with weightbearing limitations, and subject satisfaction, this research seeks to provide a more comprehensive understanding of the potential benefits of using a biofeedback device in partial weightbearing training.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years old.
* Healthy and able to walk unassisted.
* No cognitive impairments.
* Willing to participate in the study.
* Capable of using crutches.
* English- speaking.

Exclusion Criteria:

* Unwilling to participate in the study.
* Sensor incompatibility: shoe sizes smaller than EU 36 (Womens size 4, Men's size 6) or larger than EU 44 (Women's size 13, Men's size 11).
* Non-English speaking.
* Pregnant women must not take part in this study, due to a higher chance of injury in the unlikely event of a fall.
* >7 on Six-Item Cognitive Impairment Test

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Healthy subjects, aged between 18 and 60 years old able to walk unassisted.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Average peak force (Newtons, (N)) | During intervention (2-minutes)
  During partial weightbearing physical therapy routine

CONTACTS AND LOCATIONS:
Overall Officials: Justin Haller, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No